CLINICAL TRIAL: NCT05673746
Title: Acupuncture in Chemotherapy-induced Peripheral Neuropathy in Women With Breast Cancer: Acu-CIPN, a Randomized Controlled Multicenter Study
Brief Title: Acupuncture in Chemotherapy-induced Peripheral Neuropathy in Women With Breast Cancer
Acronym: Acu-CIPN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Claudio Zamagni MD, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acu-CIPN
Record Dates: First submitted 2021-05-29; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Peripheral Neuropathy
Keywords: peripheral neuropathy; breast cancer; acupuncture
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Treatment for peripheral neuropathy (including neuropathic pain), according to the standard of care (e.g. "Cetirizine", "Gabapentin"). Patient will be followed-up as per protocol for a total of 9 weeks .
  Interventions: Drug: treatment of physician choice, according to the standard of care
- Arm B (Experimental): In addition to the treatment for peripheral neuropathy and neuropathic pain, according to the standard of care (e.g. "Cetirizine", "Gabapentin"), patient will receive acupuncture administration twice a week and for a 6-week treatment period. Patient will also be followed-up for 3 weeks after the end of treatment.
  Interventions: Procedure: Acupuncture; Drug: treatment of physician choice, according to the standard of care

INTERVENTIONS:
Procedure: Acupuncture — acupuncture administration
  Arms: Arm B
Drug: treatment of physician choice, according to the standard of care — treatment of physician choice, according to the standard of care for the treatment of chemotherapy-induced peripheral neuropathy, including neuropathic pain

SUMMARY:
The main purpose of this study is to define whether acupuncture in addition to the treatment of physician choice as per standard of care leads to a greater decrease of neuropathic pain as perceived by women with breast cancer who suffer from chemotherapy-induced peripheral neuropathy. Peripheral neuropathy and neuropathic pain of hands and foots will be assessed by using a Number Rate Scale (NRS scale) and data will be compared between standard of care treatment group and acupuncture in addition to standard of care treatment group.

DETAILED DESCRIPTION:
Patients with breast cancer diagnosis and taxane-induced peripheral neuropathy since at least 1 week (CTCAE4.0 Grade 1-3 and NRS≥4) will be enrolled. Patients will be randomized 1:1 in the 2 treatment arms: treatment of physician choice as per standard of care vs acupuncture in addition to standard of care treatment. In experimental arm acupuncture will be performed twice a week for 6 weeks, for a total of 12 sessions. Peripheral neuropathy symptoms and pain at hands and foot will be recorded every day by patients by use of NRS scale. At baseline and every 3 weeks patients will complete CIPN20, EORTC QL30, SF-36 and BPI in order to compare the course of neuropathic pain and quality of life in the 2 arms.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥18 years.
* Patients with diagnosis of breast cancer (stage I-III) currently receiving taxane-based chemotherapy (paclitaxel or docetaxel) in neoadjuvant or adjuvant setting, or who have completed taxane-based chemotherapy for no more than 6 months. Concomitant treatment with trastuzumab is allowed in HER-positive patients and/or hormone therapy in patients with hormone-sensitive breast cancer.
* Chemotherapy-induced peripheral neuropathy graded 1-3, according to NCICTCAE v 4.03 criteria, for at least one week and for no more than 6 months after the completion of chemotherapy regimen.
* Neuropathic pain with ≥4 points in the numeric scale rate for at least one week
* Informed consent signed before any study-specific procedure

Exclusion Criteria:

* Patients with diagnosis of metastatic breast cancer
* Pre-existing peripheral neuropathy in the 28-day period before the start of chemotherapy
* Any pre-existing condition which can both lead to or be a concomitant factor for neuropathy onset, such as not controlled diabetes mellitus, paralysis, multiple sclerosis, AIDS and Herpes Zoster
* Patients with amputation and/or severe peripheral vascular disease (peripheral revascularization interventions needed, AOCP> stage II, rheumatologic disorders affecting arteriole or microcirculation)
* Patient with history of spinal cord surgery
* Patient with history of chronic alcoholism
* Concomitant use of pharmacological agents which can cause neuropathic pain as an adverse event, except for chemotherapy
* Patient who already experienced acupuncture for any condition
* Patient currently in treatment with duloxetine, gabapentin, pregabalin or other drugs for the treatment of neuropathic pain
* Patient with history of psychiatric disorders before breast cancer diagnosis (major depressive disorders, bipolar disorder, suicidal tendency)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of peripheral neuropathy, including neuropathic pain | 6 weeks after the start of treatment
  Reduction of peripheral neuropathy, including neuropathic pain (at least 3 points on the numeric scale rate) after the 6-week treatment period versus before the start of treatment, greater in the experimental than in the control arm.

SECONDARY OUTCOMES:
Reduction of peripheral neuropathy, including neuropathic pain | at 3 and 6 weeks after the start of treatment
  Reduction of peripheral neuropathy, including neuropathic pain (at least 3 points on the numeric scale rate) at 3 and 9 weeks after the start of treatment versus before the start of treatment, greater in the experimental than in the control arm
Improvement of peripheral neuropathy, including neuropathic pain, EORTC QLQ-CIPN20/QLQ-C30 questionnaires | at 3, 6, 9 weeks after the start of treatment
  Improvement of peripheral neuropathy, including neuropathic pain perceived by patients, assessed with EORTC QLQ-CIPN20/QLQ-C30 questionnaires, at 3, 6 and 9 weeks after the start of treatment versus before the start of treatment, greater in the experimental arm compared to the control arm.
Improvement of the quality of life, SF-36 questionnaire | 6 weeks after the start of treatment
  Improvement of the quality of life as assessed with the SF-36 questionnaire at 6 weeks after the start of treatment versus before the start of treatment, greater in the experimental arm compared to control arm.
Improvement of peripheral neuropathy, including neuropathic pain, BPI questionnaire | 6 weeks after the start of treatment
  Improvement of peripheral neuropathy, including neuropathic pain perceived by patients, assessed with BPI questionnaire, at 6 weeks after the start of treatment versus before the start of treatment, greater in the experimental arm compared to control arm.
Improvement of peripheral neuropathy, including neuropathic pain, NCICTCAE v 4.03 criteria | at 3, 6, 9 weeks after the start of treatment
  Improvement of peripheral neuropathy, including neuropathic pain evaluated by the clinician according to NCICTCAE v 4.03 criteria, at 3, 6 and 9 weeks after the start of treatment versus before the start of treatment, greater in the experimental arm compared to the control arm.
Type and frequency of adverse events occurrence due to acupuncture | at last visit, 9 weeks from start of treatment
  Comparison of the type and frequency of adverse events occurred in the two treatment arms.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliero-Universitaria di Bologna, Policlinico S. Orsola-Malpighi, SSD Oncologia Medica Addarii, Bologna
  - Fondazione Policlinico Universitario A. Gemelli IRCCS Center for Integrative Oncology, Rome

IPD SHARING:
Plan to Share IPD: No